CLINICAL TRIAL: NCT04719533
Title: Short and Long Term Outcomes of Patients With and Without Pre-marked Episiotomy Location
Brief Title: Outcomes Following Pre-marking of Episiotomy Location
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sharon Davidesko MD (Other)
Responsible Party: Sponsor-Investigator, Sharon Davidesko MD, Principal Investigator, Soroka University Medical Center
Organization: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SOR-0089-20-CTIL
Record Dates: First submitted 2020-10-02; First posted 2021-01-22 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Episiotomy; Complications; Episiotomy Extended by Laceration; Episiotomy Infection
Keywords: episiotomy; episiotomy complications; premarked episiotomy

STUDY DESIGN:
Intervention Model Description: prospective randomized-controlled trial
Who Masked: Participant
Masking Description: Patients' data recorded according to a coding system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-marked episiotomy location (Experimental): Women in this group will undergo pre-marking of episiotomy location
  Interventions: Other: Pre-marking of episiotomy location
- No pre-marked episiotomy location (No Intervention): Women in this group will not undergo pre-marking of episiotomy location

INTERVENTIONS:
Other: Pre-marking of episiotomy location — A template marking the pre-determined correct location of episiotomy will be used to mark to women in the interventional group
  Arms: Pre-marked episiotomy location

SUMMARY:
To compare short- and long-term outcomes of women following episiotomy during the second stage of labor, following marking of episiotomy location during the first stage of labor with those of women who underwent episiotomy without marking.

DETAILED DESCRIPTION:
Purpose: To compare short- and long-term outcomes of women following episiotomy during the second stage of labor, following marking of episiotomy location during the first stage of labor with those of women who underwent episiotomy without marking.

Hypothesis: Women following episiotomy following pre-marking of the location will suffer from fewer short- and long-term complications compared to those without pre-marked episiotomy location.

Study type: prospective randomized-controlled trial

ELIGIBILITY:
Inclusion Criteria:

* women 18 years of age or older who present in active labour to our center and consent to participate in the study

Exclusion Criteria:

* women under 18 years of age or those who do not or are unable to provide informed consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2025-09-24 (Estimated)

PRIMARY OUTCOMES:
Extended laceration of the episiotomy | Up to 1 hour following the episiotomy
  Additional perineal tears originating from the original episiotomy, as described in the birth chart
Third- and fourth-degree perineal tears | Up to 2 hours following the episiotomy
  Perineal tears involving the anal sphincter in addition to the episiotomy, as documented in hospital records
Post-partum hemorrhage | Up to 6 weeks following delivery
  Early (<24 hours) or later (24 hours to 6 weeks) hemorrhage following delivery requiring physician intervention as documented in medical records
Blood transfusion requirement | Up to 5 days following delivery
  Any requirement for blood products following delivery as documented in the hospital discharge
Episiotomy site infection | Up to 6 weeks following delivery
  any documented infection of the episiotomy site treated in ambulatory or hospital setting, as recorded in medical records
Requirement of resuturing of episiotomy or evacuation of hematoma | up to 6 weeks following delivery
  Any additional surgical intervention required relating to the episiotomy, as recorded in medical records
Long-term symptoms related to episiotomy | Up to 5 years following delivery
  Any symptoms including perineal pain, dyspareunia, urine incontinence or fecal incontinence as reported by women using a numerical scale or dichotomic scale where appropriate
Perineal tears in subsequent deliveries | Up to 5 years following delivery
  As recorded in hospital records
Surgical correction of episiotomy | Up to 5 years following delivery
  Any additional surgical procedures required for correction of episiotomy related symptoms as recorded in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Davidesko, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No
No data is to be shared with other researchers